CLINICAL TRIAL: NCT04276064
Title: Modulation of Sleep Perception Through Auditory Closed-loop Stimulation of Brain Oscillatory Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Nissen (Other)
Responsible Party: Sponsor-Investigator, Christoph Nissen, Chief physician, University of Bern
Organization: University of Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-02426
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Sleep; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with insomnia (Experimental): Patients with insomnia disorder according to DSM-5 criteria
  Interventions: Device: Auditory closed-loop stimulation: slow oscillation boosting; Device: Auditory closed-loop stimulation: slow oscillation disruption; Device: Sham stimulation
- Healthy controls (Experimental): Healthy controls
  Interventions: Device: Auditory closed-loop stimulation: slow oscillation boosting; Device: Auditory closed-loop stimulation: slow oscillation disruption; Device: Sham stimulation

INTERVENTIONS:
Device: Auditory closed-loop stimulation: slow oscillation boosting — Auditory-closed loop stimulation: slow oscillation boosting
Device: Auditory closed-loop stimulation: slow oscillation disruption — Auditory closed-loop stimulation: slow oscillation disruption
Device: Sham stimulation — Sham stimulation

SUMMARY:
Sleep is ubiquitous in animals and humans, and disruptions are of high clinical importance. Still, the neural basis of sleep perception is insufficiently understood, which limits the development of new treatments. The current project is designed to further contribute to the understanding of the neural basis of sleep perception and to the development of innovative treatments for disrupted sleep (insomnia).

ELIGIBILITY:
Inclusion Criteria:

* For patients: diagnosis of ID according to DSM 5 criteria; for controls: mentally and somatically healthy
* Age 18 to 65 years
* Written informed consent

Exclusion Criteria:

* Relevant current or past serious medical disorder, including but not limited to cardiac arrhythmia, diabetes mellitus, and chronic pain conditions.
* Neurological conditions including epilepsy, history of brain injury, encephalitis or any organic brain syndrome
* Current or past mental disorders (life time prevalence), e.g. depressive disorder, attention deficit disorder, psychotic disorders, anxiety disorder, posttraumatic stress disorder
* Sleep disorders (except ID for patients), including movement-related sleep disorders (PLMS index with arousal > 5) or breathing-related sleep disorders (AHI > 15)
* Intake of CNS active medication (except appropriate thyroid hormone substitution)
* Current or past substance abuse or dependency
* Smoking > 5 cigarettes per day
* Excessive caffeine consumption (> 500 mg or 5 cups coffee per day)
* Irregular sleep schedules resulting from shift work, travelling or personal habits, defined as a sleep/wake time deviation > 4 hours in the weekly routine or as a habitual total sleep time < 4.5 hours or > 10 hours per night
* Known pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Modulation Index | Averaged across NREM sleep of the baseline night (about 6 hours)
  Measure of phase-amplitude coupling

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Nissen, MD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mikutta C, Feige B, Maier JG, Hertenstein E, Holz J, Riemann D, Nissen C. Phase-amplitude coupling of sleep slow oscillatory and spindle activity correlates with overnight memory consolidation. J Sleep Res. 2019 Dec;28(6):e12835. doi: 10.1111/jsr.12835. Epub 2019 Mar 7. PMID 30848042
- See also: Website research group — https://www.upd.unibe.ch/research/research_groups/group_nissen_cooperation_univ_geneva/group_nissen_cooperation_univ_geneva/index_eng.html